CLINICAL TRIAL: NCT02702700
Title: Photo-induction as a Means to Improve Cisplatin Delivery to Pleural Malignancies: a Clinical Phase I Trial
Brief Title: Photo-induction as a Means to Improve Cisplatin Delivery to Pleural Malignancies
Acronym: PDT-lipo
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Drug supply issue
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Solange Peters, Associate physician, Centre Hospitalier Universitaire Vaudois
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUV-DO-PDT-2015
Record Dates: First submitted 2016-01-25; First posted 2016-03-09 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Pleural Effusion, Malignant
MeSH Terms: conditions — Pleural Effusion, Malignant | interventions — SPI-77, liposomal; lipoplatin; Verteporfin; Photochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lipoplatin/Visudyne-mediated photodynamic therapy (Experimental): 200 mg/m2 Lipoplatin™ will be delivered as iv perfusion. Then, intrapleural photo-induction will be realized through a classical video-assisted thoracoscopic (VATS) approach using 3 mg/m2 Visudyne® activated at 689 nm. At the end of the procedure, the patients will receive chemical pleurodesis by VATS as per standard-of-care treatment for malignant pleural effusion.
  Interventions: Drug: Cisplatin, liposomal; Drug: Verteporfin; Device: Device for Intrapleural Visudyne-mediated Low-Dose Photodynamic Therapy with integrated in situ light dosimetry

INTERVENTIONS:
Drug: Cisplatin, liposomal — Lipoplatin IV 200 mg/m2
  Other Names: Lipoplatin™
Drug: Verteporfin — Visudyne® IV 3 mg/m2
  Other Names: Visudyne®
Device: Device for Intrapleural Visudyne-mediated Low-Dose Photodynamic Therapy with integrated in situ light dosimetry — Intrapleural photo-induction will be realized in the chest cavity with low-dose PDT using Visudyne® 3mg/m2 as photosensitizer, activated by 689 nm laser light with a fluence of 10J/cm2 and a fluence rate of <10mWcm2.

SUMMARY:
This clinical study aims to explore intrapleural low-dose Visudyne®-mediated photodynamic therapy (photo-induction) as a pathway to promote the uptake of systemically administered Lipoplatin™ in pleural malignancies of patients undergoing video-assisted talcage for their malignant pleural effusions. Photo-induction is expected to overcome the chemo-resistance of pleural malignancies for cisplatin-based chemotherapeutics and thereby improve local tumor control.

DETAILED DESCRIPTION:
The primary objective of the study is to assess the safety and tolerability of intrapleural Visudyne®-mediated photo-induction as a means to selectively increase tumor uptake of systemically administered Lipoplatin™ in patients with primary or secondary pleural malignancies.

The secondary objectives are:

Assessment of treatment efficacy as measured by dyspnea reduction, pleural effusion free survival as well as local relapse rate, progression free and median overall survival.

Analysis of the pleural intratumor penetration of Lipoplatin™ by repeated biopsies for Lipoplatin concentration measurements before and after Visudyne® treatment as well as vessel modulation related parameters (pericyte coverage, vessels morphology).

ELIGIBILITY:
Inclusion criteria

* Stage IV breast, ovarian, gastric, colorectal, germ cell, lung, bladder, sarcoma or head and neck carcinoma requiring systemic chemotherapy OR alternatively
* Stage I/II malignant pleural mesothelioma OR alternatively
* Stage III/IV mesothelioma requiring systemic chemotherapy OR alternatively
* Stage IVa thymic malignancies AND
* Cytologically proven malignant pleural effusion requiring VATS pleurodesis
* PS 0-1
* Age 18-80
* Written informed content
* Life expectancy >3 months
* Laboratory Requirements - within 28 days prior to enrollment:
* Haematology:

  * absolute granulocytes ≥1× 109/L
  * platelets ≥100 × 109/L
  * leukocytes ≥3 × 109
* Biochemistry:

  * Bilirubin ≤3 × upper limit of normal (<5x if liver metastasis present)
  * AST(SGOT) ≤2.5 × upper limit of normal (<5x if liver metastasis present)
  * Creatinine clearance ≥50 mL/min according to Cockroft and Gault
* No major cardio-pulmonary co-morbidity precluding a surgical approach according to local standards
* Enrollment decision at the institutional multidisciplinary tumor board
* Patient must be willing to use effective methods of contraception. Female patients must be postmenopausal, surgically sterile, or they must agree to use a physical barrier method of contraception in addition to either an intrauterine device or hormonal contraception until at least of 3 months after the study treatment. Male patients must agree to use a barrier method (condom) for 3 months after study treatment.

Exclusion criteria

* Grade >2 peripheral neuropathy
* Any concurrent anticancer systemic therapy within 14 days before the study intervention
* Any condition that is unstable or could jeopardize the safety of the patient and their compliance in the study e.g. Known or suspected allergy to the investigational agent or any agent given in association with this trial.

Clinically serious infections requiring systemic antibiotic (e.g antiviral, antimicrobial, antifungal) therapy.

* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Severe interstitial pneumonia or pulmonary fibrosis
* Chronic corticosteroid use at equivalent dose of >30mg/d methylprednisolone
* Pregnancy or breast-feeding
* Porphyria
* Severe liver insufficiency

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-01; Primary Completion 2018-08-28 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
Safety of the treatment as assessed by 30-day postoperative mortality | 30 days
  survival status at 30 days
Tolerability of the treatment as assessed by 30-day postoperative mortality | 30 days
  survival status at 30 days
Feasibility | 30 days
  survival status at 30 days
Acute respiratory failure rate | 30-day postoperative
Dyspnea according to CTCAE v4.0 | 30-day postoperative
Chest pain rate according to CTCAE v4.0 | 30-day postoperative
Dyspnea according to Medical Research Council (MRC) chronic dyspnea scale (5-point) | 30-day postoperative

SECONDARY OUTCOMES:
Malignant effusion recurrence-free - percentage of patients without recurrent pleural effusion at 30 days | 30 days after treatment
Dyspnea reduction according to CTCAE v4.0 | 30 days after treatment
  CTCAE v4.0
Tumor response | according to local standard
  Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Overall survival (OS) | every 3 months up to 3 years
Overall response rate (ORR) based on investigator assessment according to Response | according to local standard
  Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Progression-free survival (PFS) | according to local standard
  Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Duration of Response (DOR) | according to local standard
  Evaluation Criteria in Solid Tumors (RECIST) version 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Beat Ris, MD, Prof., Study Director — CHUV
Locations (1):
- Oncology Department, Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Vaud (VD), Switzerland